CLINICAL TRIAL: NCT00198302
Title: A Phase II, Randomized, Double-blind, Multi-center Clinical Trial Comparing Safety and Pharmacokinetics of Standard Antibiotic Therapy, Plus Aurexis® or Placebo, for Treatment of Staphylococcus Aureus Bacteremia (SAB)
Brief Title: Clinical Trial Comparing Safety and Pharmacokinetics of Standard Antibiotic Therapy, Plus Aurexis® or Placebo, for Treatment of Staphylococcus Aureus Bacteremia (SAB)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: INH-AUR-002
Record Dates: First submitted 2005-09-09; First posted 2005-09-20 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Staphylococcus Aureus Bacteremia
Keywords: staphylococcus aureus; bacteremia; sepsis
MeSH Terms: conditions — Staphylococcal Infections; Bacteremia; Sepsis

INTERVENTIONS:
Drug: Aurexis®

SUMMARY:
Hospitalized patients at least 18 years of age, with Staphylococcus aureus bacteremia (SAB) will be enrolled into the study and receive one dose of Aurexis® intravenously on Study Day 1, and will be followed until Study Day 57. Aurexis is a humanized monoclonal antibody that is designed to combat Staphylococcus aureus.

The purpose of this study is to assess the safety and pharmacokinetics of standard antibiotic therapy, plus Aurexis or Placebo for treatment of (SAB). Additionally, certain tests and measurements will be conducted to preliminarily determine if Aurexis demonstrates any benefit to these patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 18 years old
* Informed consent obtained from subject or legal guardian
* Willing to practice reliable birth control measures during the study period
* Diagnosis of SAB, as evidenced by clinical symptoms and one positive blood culture obtained ≤ 72 hours prior to initiation of study drug infusion

Exclusion Criteria:

* Pregnant or nursing females
* Polymicrobial bacteremia
* Diagnosis of septic shock (refer to APPENDIX B)
* Neutropenia (absolute neutrophil count < 500/mm³)
* Undergoing any type of dialysis or expected to start dialysis within 30 days
* Moribund clinical condition with a high likelihood of death within 72 hours of randomization
* Received an investigational drug within 30 days of study entry
* Considered unlikely to comply with the study procedures or to return for scheduled post-treatment evaluations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Study Completion 2005-02

PRIMARY OUTCOMES:
• To evaluate the safety of standard of care, plus a single dose of Aurexis® compared to a single dose of placebo, in subjects with documented SAB
• To evaluate the pharmacokinetics of a single dose of Aurexis® in combination with standard of care in the subjects with SAB
• To evaluate the activity of a single dose of Aurexis® in combination with standard of care, as measured by:
o number of subjects with uncomplicated SAB at baseline who progress to complicated SAB
o number of subjects with microbiologically documented relapse of SAB
o mortality rates

SECONDARY OUTCOMES:
• To evaluate the effect of a single dose of Aurexis® in combination with standard of care on the:
o proportion of subjects who develop sepsis, severe sepsis, or septic shock
o time to achieve a negative blood culture
o time to defervescence
o mean (and median) number of days in the hospital and ICU
o mean (and median) number of days requiring mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Seth Hetherington, M.D., Study Director — Inhibitex